CLINICAL TRIAL: NCT07369245
Title: Randomized Controlled Trial to Evaluate the Efficacy of Hypnosis and Learning Self-exercises for Outpatients With Moderate to Severe Alcohol Addiction
Brief Title: Techniques for Activating Consciousness (TAC) for Outpatients With Moderate to Severe Alcohol Addiction
Acronym: TAC-ADDICT
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Versailles Hospital (Other)
Responsible Party: Principal Investigator, Dr Claire FARINA, Investigator Coordonnator, Versailles Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: P23/03 - TAC-ADDICT
Record Dates: First submitted 2025-12-30; First posted 2026-01-27 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2025-11

CONDITIONS: Alcohol Addiction
Keywords: Hypnotic therapy; Techniques for Activating Consciousness (TAC); Alcohol addiction
MeSH Terms: conditions — Alcoholism

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention)
- TAC intervention (Experimental)
  Interventions: Behavioral: TAC intervention

INTERVENTIONS:
Behavioral: TAC intervention — Patients receiving TAC (Techniques for Activating Consciousness) intervention in addition to standard care
  Arms: TAC intervention

SUMMARY:
Many patients are considering the use of so-called "hypnosis" treatments in the field of addictions. However, these techniques lack sufficient levels of evidence with regard to the standards required by Evidence-Based Medicine.

In other domains, however, hypnosis has demonstrated an interesting level of evidence, particularly in pain management.

The investigators will focus on the "Techniques for Activating Consciousness" (TAC), which represent an optimized therapeutic approach derived from hypnotic therapy.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients consulting for an alcohol-related addiction problem at the CSAPA of Versailles (sites in Versailles, Trappes, Rambouillet) or at the Centre Hospitalier des 4 Villes (day hospital or CSAPA in Sèvres)
* Patients must meet at least 4 of the 11 DSM-5 criteria (Annex 2), corresponding to moderate to severe addiction
* Patients must be affiliated with the French social security system

Exclusion Criteria:

* Refusal to participate
* Decompensated psychiatric pathology contraindicating therapy:

  * Presence at inclusion of delusional, dissociative, and/or persecutory symptoms
  * Presence at inclusion of hypomanic or manic decompensation
* Severe cognitive impairment, evidenced by inability to perform the clock-drawing test (draw the clock face, place the numbers, and set the hands to 11:10)
* Adults legally protected under French law (deprivation of liberty, legal safeguard, guardianship, curatorship)
* Inability to understand French

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 98 (Estimated)
Dates: Start 2026-01-15 (Estimated); Primary Completion 2027-07-15 (Estimated); Study Completion 2028-01-15 (Estimated)

PRIMARY OUTCOMES:
The patient's ability to control alcohol consumption during outpatient follow-up in a CSAPA | 6 months
  The main outcome measure will be the number of weeks to achieve the targeted goal between T0 (first consultation when the objective is set) and M6 (cumulative time).

SECONDARY OUTCOMES:
Controlling addictive behavior in both groups | 12 months
  Evaluation criteria for both groups:
  * Cumulative time over 12 months during which the subject meets the target of controlling addictive behavior; percentage of time at target between T0-M6 and T0-M12; number of weeks to reach the target; number of relapses between T0-M6 and T0-M12; time between achieving the target and relapse between T0-M12
  * Craving intensity (weekly via electronic patient questionnaire)
  * Levels of anxiety and depression (HAD scale) and global relaxation (IERS-3), at T0, M6, and M12
  * Care received (interventions, medications) from medical records at M6 and M12
  * Patient opinion questionnaire at M6 and M12 on what was perceived as useful or not in their treatment
Evaluation criteria for the TAC group | 12 months
  Weekly self-reports (via electronic patient questionnaire) on the frequency of exercise practice, perceived effectiveness of TAC (Techniques for Activating Consciousness) on their addictive issues (VAS 0-10), and tolerance of TAC (Techniques for Activating Consciousness)

CONTACTS AND LOCATIONS:
Locations (2):
- France (2):
  - Hospital Versailles, Le Chesnay
  - CH des 4 Villes, Sèvres